CLINICAL TRIAL: NCT06282315
Title: A Pragmatic Phase III Multicentre Clinical Trial to Evaluate the Safety and Effectiveness of a Single Dose of an Albendazole-Ivermectin Coformulation vs Albendazole for Preventive Chemotherapy of Soil-Transmitted Helminth Infections in School-Aged Children
Brief Title: Real World Evaluation of an Albendazole-Ivermectin Coformulation Safety and Effectiveness
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Insud Pharma (Industry)
Collaborators: Ghana Health Services (Other Government); Kenya Medical Research Institute (Other); Bridges to Development (Unknown); Sanger Institute (Unknown); Barcelona Institute for Global Health (Other); European Union (Other); Swiss Confederation (Unknown); Fundación Mundo Sano (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REALISE
Record Dates: First submitted 2024-02-06; First posted 2024-02-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Soil-Transmitted Helminths
Keywords: STH; albendazole; ivermectin; hookworms
MeSH Terms: conditions — Hookworm Infections | interventions — Random Allocation; Mass Drug Administration; Watchful Waiting

STUDY DESIGN:
Intervention Model Description: Open-label, randomized at the school level, and each eligible participant within a school will receive only one of the study treatments (ALB or IVM+ALB).
Who Masked: Outcomes Assessor
Masking Description: This is an open study. Participants and the study investigators assessing drug safety will not be blinded to treatment arms. Only the laboratory-based effectiveness measurement will be performed by blinded operators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed Dose Combination (FDC) albendazole and Ivermectin (ALB/IVM ) (Experimental): Single dose of a tablet of FDC 400 mg/18 mg IVM or 400 mg ALB/9 mg IVM, administered according to the following age criteria:
  1. For children from 5-14 years old (included) at the time of screening visit: 1 tablet of FDC 400 mg ALB/9 mg IVM
  2. For children from 15-17 years old (included) at the time of screening visit: 1 tablet of FDC 400 mg ALB/18 mg IVM
  Interventions: Drug: Pre-screening Phase; Drug: Screenig Phase; Drug: Randomization; Drug: Baseline Effectiveness Cohort; Drug: Day 0 Trial Intervention; Drug: Active Surveillance (study visit Day 1, Day 2 and Day 7); Drug: Passive Surveillance; Drug: Post-Treatment Effectiveness Evaluation
- Albendazole (ALB) (Active Comparator): Single dose of a tablet of ALB 400 mg (active control arm).
  Interventions: Drug: Pre-screening Phase; Drug: Screenig Phase; Drug: Randomization; Drug: Baseline Effectiveness Cohort; Drug: Day 0 Trial Intervention; Drug: Active Surveillance (study visit Day 1, Day 2 and Day 7); Drug: Passive Surveillance; Drug: Post-Treatment Effectiveness Evaluation

INTERVENTIONS:
Drug: Pre-screening Phase — The entire school population will be invited to participate in the study. The purpose of this phase is to confirm participant eligibility for enrolment in the study based on the inclusion and exclusion criteria. Given the context in which the clinical trial is being conducted, in many instances, group meetings with the parents/guardians of potential participants in the community or at school might be necessary as part of the informed consent process. This consent process may be performed up to three months before the start of the screening visit activities.
  Participants and parents/guardians of subjects will be asked to confirm in writing their agreement to participate in the trial before any study-specific procedure is conducted. In addition, written assent will be sought for participants over 12 years of age.
Drug: Screenig Phase — The purpose of the screening visit is to confirm subject eligibility for enrolment in the study based on the inclusion/exclusion criteria. Screening visits in a particular school can be performed between 14 and 7 days before the intervention (Day 0).
  To continue with the screening activities, participants must have signed written consent from their parent or legal guardian, and in the case of participants aged 12 years or older, they must also have a signed assent form before any specific study procedure is performed.If the consent/assent process has not been finalized during the pre-screening phase, this can be completed during the screening visit, but always before any trial procedure.
  All participants who consent to participate in the trial will be given a Participant Screening Number, which will be assigned sequentially as the informed and assent forms are signed.
Drug: Randomization — Only when the screening process is finalized in a particular school, and the list of eligible participants is closed, with at least 100 eligible participants, will the school be a candidate for randomization. Once the screening process is finalized, the investigator or designee will notify the ISGlobal Trial Statistician, who will provide the School Randomization ID allocated based on the randomization lists created before the trial starts. School Randomization ID will be assigned sequentially per site, following the order of school randomization. Additionally, the ISGlobal Trial Statistician will provide the site with the list of eligible participants per school randomly selected to participate in the Effectiveness Cohort.
Drug: Baseline Effectiveness Cohort — Before the administration of the study drug at school, participants selected for the Effectiveness Cohort will perform an additional study visit during which they will provide the study team with a stool sample for STH analysis. A dried blood spot (DBS) sample will also be taken to test for S. stercoralis.
  Sampling of the baseline effectiveness cohort will be conducted within 7 days before the start of the school study intervention. In addition to the delivery of the stool/blood sample, participants from the effectiveness cohort will be evaluated for scabies by designated study personnel following the IACs simplified criteria.
Drug: Day 0 Trial Intervention — Within seven days after the first sample for the baseline effectiveness cohort is collected, the school's mass administration of the allocated drug will take place. All participants included in the list of eligible subjects from a particular randomized school will receive a single dose of the medication administered to their school (FDC or ALB). Before the administration, participants will be asked about any medical condition that has arisen since the last study visit, in which case information will be documented as a concomitant disease.
  In case a participant vomits within one hour after the study drug intake (during the study physician observation period), the participant will continue participating in the trial and may still participate in the effectiveness cohort. If they are chosen for the day 21 or month 11 effectiveness cohort, an additional sensitivity analysis will be performed without including these participants, considered as Intervention Fail.
  Other Names: Mass Drug Administration (MDA)
Drug: Active Surveillance (study visit Day 1, Day 2 and Day 7) — Active safety surveillance will be performed at school during the trial intervention on day 0 until day 7 post-intervention. The assessment will include recording of all AEs and SAEs presented by study participants from the intake of the study drugs, and for two additional days (Day 1 and Day 2 study visits). During active surveillance, participants will be visited by a study physician at school during the study intervention, on day one and day two, and they will be questioned about any potential AE or change in a pre-existing condition. In addition, a final safety visit will be conducted to all participants at Day 7 to collect data on any potential AE occurred between day 2 and the end of the surveillance period and to perform a follow up of any AE ongoing after Day 2 visit.
Drug: Passive Surveillance — Passive surveillance will be carried out by monitoring AEs in health facilities near the schools involved in the study for six days after the intervention until Day 7 (end of the safety surveillance period). Although AE will be actively monitored during the scheduled study visits, this passive surveillance will allow for the identification of AEs and potential SAEs that might occur and remained underreported in case the participant does not attend school during the active safety surveillance period. In addition, a diary cards will be given to participants to write any AE they may have from Day 2 to Day 6 post intervention.
Drug: Post-Treatment Effectiveness Evaluation — Post-treatment effectiveness evaluation will be performed by measuring the prevalence of STH at two time points: 21 days after the intervention (± 7 days) and 11 months after intervention (± 28 days). Additionally, the reduction in S. stercoralis seroprevalence will be evaluated 11 months after the intervention.
  These participants will be tested for STH by Kato-Katz at the two post-treatment time points (day 21 and month 11) and for S. stercoralis by NIE ELISA at 11 months. The diagnostic test will be the same as in the intervention of Baseline Effectiveness Cohort.
  As part of the genetic monitoring pilot study and the microbiome analysis, the same samples will be collected as described in the intervection of Baseline Effectiveness Cohort.

SUMMARY:
An open-label, randomized by school, two-arm pragmatic trial, will be conducted involving two study sites in Sub-Saharan-Africa (SSA), Ghana and Kenya, to evaluate safety and effectiveness of the newly developed fixed dose combination (FDC) of albendazole (ALB) and ivermectin (IVM) as a single dose to treat Soil-Transmitted Helminths (STH), compared to the standard dose ALB single dose for the treatment and control of STH (REALISE study: Real World Evaluation of an Albendazole-Ivermectin Coformulation Safety and Effectiveness). The general objectives are to validate the benefits of FDC through this pragmatic trial in a context of mass drug administration (MDA) programme to evaluate the safety as a primary endpoint and effectiveness profile as a secondary endpoint, in a large population of school-aged children.

DETAILED DESCRIPTION:
In the REALISE study a total of 20,000 children will be enrolled approximately in both countries for the safety cohort, 10,000 children in around 30 schools per country (5,000 per treatment arm). For the effectiveness cohort, REALISE study is planned to assess a total of approximately 4,500 participants in both countries, 2,250 children per country (75 children for each of the 30 schools and 1,125 children per treatment arm).

The REALISE study will have two study arms:

* Treatment arm 1: Single dose of a tablet of FDC 400 mg/18 mg IVM or 400 mg ALB/9 mg IVM, administered according to the following age criteria:

  1. For children from 5-14 years old (included) at the time of screening visit: 1 tablet of FDC 400 mg ALB/9 mg IVM.
  2. For children from 15-17 years old (included) at the time of screening visit: 1 tablet of FDC 400 mg ALB/18 mg IVM.
* Treatment arm 2: Single dose of a tablet of ALB 400 mg (active control arm).

Randomization will occur at the school level, and each eligible participant within a school will receive only one of the study treatments. Given the variable number of children in the Ghanaian and Kenyan schools, and that conducting the intervention for only a fraction of the school is not feasible, it may be possible to exceed the intended trial sample size. Efforts will be made to minimize this

The Primary objective of the trial will be to evaluate and compare safety of a FDC against ALB alone via MDA in two study areas in Kenya and Ghana in the seven days after first treatment intervention. Thus, as a primary outcome, the adverse effects will be monitored through a specific surveillance system established in schools, hospitals and health centers as health facilities. Safety surveillance will be performed for seven days after each MDA, allowing for the identification of AEs and SAEs in subpopulations (in terms of gender, age, body weight, comorbidities, and additional risk factors) for better estimation of safety.

This surveillance will consist of active surveillance at day 0, day 1, day 2 and day 7 post-intervention to record any AEs and SAEs presented by participants during the conducting study with drug intake. In addition, the trial will include passive surveillance monitoring AEs and SAEs through diary cards given to the subjects, and in hospitals and health centres near the schools involved in the study for six days after the intervention until day 7 (end of the safety surveillance period) to avoid the loss of possible AEs and SAEs underreported, in case the participant does not attend school during the surveillance period.

The Secondary objective will be to evaluate the effectiveness of one round of MDA with FDC compared to ALB against STH T. trichiura by microscopy, to address the reduction of the prevalence of this species in the FDC and ALB arms. Thus, the secondary outcome will be measured at the school level, prior to the first intervention (baseline), at 21 days post intervention and within the month prior to the second yearly intervention which is at s11 months.

Moreover, the trial will include Exploratory objectives to evaluate the effectiveness of one round of MDA with FDC compared to ALB against S. Stercolaris by serology to address the outcome of the seroprevalence reduction of this species in the FDC arm and ALB arm and to evaluate the effectiveness of one round of MDA with FDC compared with ALB against Hookworms and A. lumbricoides to determine the reduction of the prevalence of these species through microscopy.

The frequency of scabies also will be measured as an exploratory objective in the effectiveness cohort at baseline and 21 days after the intervention.

Genetic monitoring is an exploratory objective to address the impact of the two treatment arms on the genetic structure of the populations of parasites. This genetic analysis will measure on the one hand the genetic diversity as an estimation of the effective population size and a proxy for successful control programmes, as seen for other parasites (it is expected that diversity will be lower in populations closed to elimination. In addition, the genetic differentiation between baseline parasites and the parasites collected after the interventions will be evaluated. Thus, the investigators will be able to evaluate the impact of both treatments in genetic selection and potentially identify genes associated with treatment failure and anthelmintic resistance. On the other hand, the investigators will measure the genome-wide association to see the relationship between parasite genetics and parasite clearance in response to treatments.

As part of the exploratory endpoints, the investigators will estimate alpha and beta diversity as well as the composition of the microbiome at phylum, family and genus level for each sample and time point. Investigators will assess differences between infected and uninfected participants at baseline by comparing the diversity and relative abundance of the different bacteria between baseline and 21 days after the intervention, comparing the effect of the two treatment arms in the microbiome composition. Moreover, the investigators will also explore the recovering of the initial microbiome composition between month 11 post-intervention and baseline, particularly in those participants that were not newly infected after 11 months.

ELIGIBILITY:
Inclusion Criteria:

Individuals of both sexes that attend the selected schools in the trial areas in Ghana and Kenya that meet the following criteria:

1. Age: 5 to 17 years old (included).
2. Height: over 110 cm.
3. Parental acceptance to participate in the study by obtaining written informed consent approved by the Ethics Committee. Written assent will also be obtained from children according to the local national legislation (12-17 years old).

   Exclusion Criteria:
4. Epidemiological risk of being infected by Loa loa, defined as those who have visited any of the following countries: Angola, Cameroon, Central Africa Republic, Chad, Congo, Democratic Republic of the Congo, Equatorial Guinea, Ethiopia, Gabon, Nigeria and Sudan.
5. Serious medical illness, defined as participants showing symptoms of acute illness which could hamper the participation in the trial, such as high-grade fever, severe diarrhoea, neurological symptoms or others, per investigator's criteria.
6. Any condition prevents the appropriate evaluation and follow-up of the participant, per the investigator's criteria.
7. Known hypersensitivity to any component of either study treatment.
8. Pregnant or first week post-partum: female participants who are post-menarche must have a negative urine pregnancy test at screening.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
AEs and SAEs record of participants treated with FDC compared to ALB. | 7 days, active surveillance (Day 0 (1 hour), Day 1, Day 2 and Day 7 post-intervention) and passive surveillance (From Day 0 up to Day 6 post-intervention)
  Adverse events will be recorded in the source documents and the electronic Case Report Form during the trial. The nature of the AE, its date and time of onset, duration and severity, therapy employed (only for SAEs) and the investigator's opinion of causality to the study drug with an alternate aetiology, if appropriate, will be documented.
  Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of intensity.
  Classification of the AEs and SAEs according to their frequency will be performed by the Sponsor at the end of the trial.

SECONDARY OUTCOMES:
Reduction in T. trichiura prevalence in participants treated with FDC compared with ALB. | Baseline, 21 days and 11 months post-intervention
  At each time point, one stool sample will be requested from each selected participant, and the presence and number of STH eggs will be determined by a single Kato Katz method (WHO gold standard for STH diagnosis) using microscopy. T. trichiura prevalence will be considered as the number of participants infected divided by the total number of participants in the effectiveness cohort.
  STH diagnosis by Kato-Katz on fresh stool (samples analysed up to a maximum of 24 hours after sample collection). The stool sample will be analysed in the local laboratory to estimate STH prevalence at baseline in each school as part of evaluating the STH effectiveness of the treatment arms.

OTHER OUTCOMES:
Exploratory 1: Reduction in Strongyloides stercoralis seroprevalence in participants treated with FDC compared with ALB. | Baseline and 11 months
  A dried blood spot (DBS) will be obtained from the selected effectiveness cohort at each time point. The presence of specific antibodies against S. stercoralis will be determined by standard serology methods (ELISA). The seroprevalence of S. stercoralis will be calculated as the number of participants with a positive result by serology divided by the total number of participants in the effectiveness cohort.
  For the ELISA assay based on the recombinant S. stercoralis NIE antigen, a few drops of blood will be taken from the participants using Dried blood spot testing (DBS) to estimate the baseline prevalence of S. stercoralis.
Exploratory 2: Reduction in hookworms prevalence in participants treated with FDC compared with ALB. | Baseline, 21 days and 11 months post-intervention
  At each time point, one stool sample will be requested from each selected participant, and the presence and number of STH eggs will be determined by a single Kato Katz method (WHO gold standard for STH diagnosis) using microscopy. Hookworms prevalence will be considered as the number of participants infected and divided by the total number of participants in the effectiveness cohort.
  STH diagnosis by Kato-Katz on fresh stool (samples analysed up to a maximum of 24 hours after sample collection). The stool sample will be analysed in the local laboratory to estimate STH prevalence at baseline in each school as part of evaluating the STH effectiveness of the treatment arms.
Exploratory 3: Reduction in A. lumbricoides prevalence in participants treated with FDC compared with ALB. | Baseline, 21 days and 11 months post-intervention
  At each time point, one stool sample will be requested from each selected participant, and the presence and number of STH eggs will be determined by a single Kato Katz method (WHO gold standard for STH diagnosis) using microscopy. A.lumbricoides prevalence will be considered as the number of participants infected and divided by the total number of participants in the effectiveness cohort.
  STH diagnosis by Kato-Katz on fresh stool (samples analysed up to a maximum of 24 hours after sample collection). The stool sample will be analysed in the local laboratory to estimate STH prevalence at baseline in each school as part of evaluating the STH effectiveness of the treatment arms.
Exploratory 4: Describe the frequency of scabies before and after the intervention in the two treatment arms. | Baseline and 21days
  Frequency of scabies measured by IACS simplified criteria. The frequency of scabies will be calculated as the number of participants infected divided by the total number of participants in the effectiveness cohort.
Exploratory 5: (i) Genetic diversity within and between T. trichiura populations, relative to the FDC or ALB study participants. | Baseline and 11 months
  STH positive faecal samples collected from the effectiveness cohort will undergo egg concentration, DNA extraction and whole genome sequencing.Three and a half grams or 5ml of stool from all positive samples will be stored in each study site at -80ºC before shipment to the Wellcome Sanger Institute (WSI). Libraries will be sequenced using 150 bp paired-end chemistry on an Illumina NovaSeq platform.
  Genetic diversity (measured as nucleotide diversity (pi), Watson estimator, Tajima's D) will be measured as an estimation of the effective population size and a proxy for successful control programmes, as seen for other parasites (it is expected that diversity will be lower in populations closed to elimination). In addition, the genetic differentiation (Fst) between baseline parasites and the parasites collected after the interventions will be evaluated to potentially identify genes associated with treatment failure and anthelmintic resistance.
Exploratory 5: (ii) Genetic diversity in candidate genes and identification of genes and/or regions in the genome of T. trichiura under selective pressure due to the treatment with FDC and/or ALB; | Baseline and 11 months
  STH positive faecal samples collected as indicated in (i).
  The relationship between parasite genetics and parasite clearance in response to treatment will be tested by performing genome-wide association between groups of samples 'good clearance' phenotypes (defined as a decrease in egg counts, and/or a decrease in genetic diversity over treatment time) and post interventions samples from children with poor clearance phenotypes (abnormal egg counts and/or genetic diversity over treatment time). Other variables will be included as potential confounders, such as sex, age, school and/or community. Finally, the association of beta-tubulin gene variants and resistance in the context of variants identified in the genome-wide analyses will be assessed. Once resistant parasite populations are identified, the impact of the two treatment strategies in selecting resistant strains can be evaluated.
Exploratory 5: (iii) Relative abundance of mixed parasite species within and between populations and in response to treatment in the FDC or ALB study participants. | Baseline and 11 months
  STH positive faecal samples collected from the effectiveness cohort will undergo egg concentration, DNA extraction and whole genome sequencing.
  Three and a half grams or 5ml of stool from all positive samples will be stored in each study site at -80ºC before shipment to the Wellcome Sanger Institute (WSI). Then DNA extraction will be carried out using a previously validated, highly efficient DNA extraction method for T. trichiura. DNA sequencing libraries will be prepared following established protocols by the sample management team at the WSI. Libraries will be sequenced using 150 bp paired-end chemistry on an Illumina NovaSeq platform.
Exploratory 6: (i) Characterization of the microbiome composition at baseline and its implication in MDA effectiveness | Baseline
  The microbiome composition (defined as alpha and beta diversity, as well as composition of bacteria) of stool samples collected from school aged children at baseline will be characterised. This information will be used to assess the differences between and within countries, as well as to explore if the microbiome composition can be used to predict the MDA effectiveness at cluster level.
  Two grams of stool from all participants will be stored at -80ºC before shipment to the WSI for microbiome analysis. Once at WSI, a standard validated pipeline for shotgun metagenomic sequencing will be applied on all selected samples to characterise the microbiome composition.
Exploratory 6: (ii) Determine the Impact of MDA with ALB or FDC on the microbiome composition at population level | 21 days post-treatment
  The investigators will also study the microbiome 21 days post-treatment to evaluate the impact of the two different treatment arms on the microbiome composition (defined as alpha and beta diversity, as well as composition of bacteria), as well as the potential role of the microbiome in the reinfection with STH.
  Two grams of stool from all participants will be stored at -80ºC before shipment to the WSI for microbiome analysis. Once at WSI, a standard validated pipeline for shotgun metagenomic sequencing will be applied on all selected samples to characterise the microbiome composition.
Exploratory 6: (iii) Measure the Recovery of the baseline microbiome composition at 11 months post-treatment and its role in reinfection with STH. | 11 months post-treatment
  Finally, investigators will explore the recovery of the original microbiome composition (defined as alpha and beta diversity, as well as composition of bacteria) by characterizing the microbiome on month 11 post-intervention. In addition, we will assess the differences in the microbiomes between infected and uninfected participants, subsequently stratifying by STH species and timepoint.
  Two grams of stool from all participants will be stored at -80ºC before shipment to the WSI for microbiome analysis. Once at WSI, a standard validated pipeline for shotgun metagenomic sequencing will be applied on all selected samples to characterise the microbiome composition.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Krolewiecki, MD, Principal Investigator — Insud Pharma
Locations (2):
- Ghana Health Service (GHS), Accra, Accra, Ghana
- Kenya Medical Research Institution (KEMRI), Nairobi, Nairobi County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://stop2030.org/